CLINICAL TRIAL: NCT02880410
Title: Feasibility Study on Laser Interstitial Thermal Therapy Ablation for the Treatment of Newly Diagnosed Glioblastoma
Brief Title: Feasibility Study on LITT for Newly Diagnosed Glioblastoma
Acronym: FLAG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated (failure to enroll)
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLAG
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2021-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; NeuroBlate; LITT; Quality of Life
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- LITT Treatment w/radiation therapy and temozolomide (Experimental): This is a single arm study. All eligible study subjects will undergo LITT with the NeuroBlate System in combination with radiation therapy and temozolomide
  Interventions: Device: NeuroBlate System; Drug: Radiation therapy and temozolomide

INTERVENTIONS:
Device: NeuroBlate System — Laser Interstitial Thermal Therapy
Drug: Radiation therapy and temozolomide — Radiation therapy and temozolomide

SUMMARY:
Multicenter, open-label, prospective designed study to characterize the performance of brain laser interstitial thermal therapy (LITT) ablation using the Monteris NeuroBlate System in combination with standard of care radiation therapy and temozolomide for the treatment of newly diagnosed glioblastomas (GBM).

ELIGIBILITY:
Relevant Inclusion Criteria:

1. Biopsy proven supratentorial GBM that has not undergone previous surgical resection, radiation and/or chemotherapy
2. Single enhancing lesion that is >1 cm, but < 4 cm in cross-sectional dimension, including thalamic tumor (≤ 3 cm)
3. The patient must be ≥18 years of age
4. KPS > 70
5. Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder. Patients with prior malignancies must be disease-free for five years.
6. Stable cardiovascular, pulmonary health status

Relevant Exclusion Criteria:

1. Seizures occurrence or the requirement of escalation (or addition) of anti-epileptic drugs
2. Symptoms due to mass effect of the tumor including high intracranial pressure, marked edema or ≥5mm midline shift significant
3. Uncontrolled cardiovascular conditions of hypertension (systolic >180 mm Hg), angina pectoris, or cardiac dysrhythmia; or recent history of intracranial hemorrhage
4. Serious infection, immunosuppression or concurrent medical condition (chronic or acute in nature) that may prevent safe participation or ability to meet follow-up requirements
5. Pregnancy, or planning to become pregnant
6. Patients whose physical dimensions cannot be accommodated in the MRI scanner or patients with contraindications to MRI imaging such as pacemakers, non-compatible aneurysm clips, shrapnel and other internal ferromagnetic objects
7. Patients with multiple or multifocal GBM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 2 Years
  Characterize adverse events experienced in glioblastoma subjects undergoing LITT using the NeuroBlate System. Adverse events will be collected based on subject reports and subject examination/testing.

SECONDARY OUTCOMES:
Progression-Free Survival Rate | 2 Years
  To describe progression-free survival rate in subjects with newly diagnosed glioblastomas treated with the NeuroBlate System
Overall Survival | 2 Years
  To describe/estimate the overall survival of subjects with newly diagnosed glioblastomas treated with LITT using the NeuroBlate System
Changes in Quality of Life | 2 Years
  Characterize the changes in quality of life in subjects with newly diagnosed glioblastoma who are undergoing LITT using the NeuroBlate System via Quality of Life and neurocognitive assessment tools

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, MD, Principal Investigator — The Cleveland Clinic; Sujit Prabhu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Washington University, St Louis, Missouri
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas